CLINICAL TRIAL: NCT01885039
Title: Characterization of Molecular Subtypes of Breast Cancer and Their Relationships With Known Breast Cancer Risk Factors Among Chinese Women in Hong Kong - A Pilot Study
Brief Title: Breast Tissue Study of Breast Diseases Among Women in Hong Kong
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913137; 13-C-N137
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: Cancer; Breast Cancer; Molecular Subtypes; Asian Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biospecimens: Fresh frozen and fixed tissues (breast tumor and adjacent normal tissue)

SUMMARY:
Background:

- The Chinese University of Hong Kong and the National Cancer Institute are conducting a breast tissue study in connection with another study on breast health. This larger study will look at breast health in women who live in Hong Kong. Women in the breast health study will provide a breast tissue sample during biopsy surgery. Researchers want to use part of the sample to study changes in breast tissue that are related to breast diseases. This sample study is part of the larger study.

Objectives:

- To look at changes in breast tissue that are related to breast diseases.

Eligibility:

* Women who are participating in the Hong Kong breast health study.
* Participants must be having a biopsy to remove breast tissue for study.

Design:

* Participants will have a biopsy to remove a breast tissue sample. Most of the sample will be used for diagnosis. A portion of the leftover tissue will be used for this study.
* No extra surgery will be required.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Background: Breast cancer incidence is increasing rapidly among many Asian populations primarily due to the adaptation of a Westernized lifestyle. However, Asian women seem to have a distinctive profile of breast cancer that differs from that seen in Western populations, such as earlier age at onset, more advanced stage, and higher frequency of ER-negative tumors. The disproportionally high rates among younger women were also seen among U.S.-born Asian women, such as Chinese, Filipina, Indian, and Pakistani women. These findings suggest that Asian breast cancer may have a distinct etiology that is not fully explained by adapting a westernized lifestyle. Recent molecular studies have suggested that breast cancers comprise several biologically and clinically distinct tumor subtypes. Epidemiologic evidence suggests that associations with breast cancer risk factors may vary by tumor subtype. However, most previous studies were conducted in Western populations; large, population-based epidemiologic studies characterizing molecular subtypes of breast cancer in Asian women are limited. In this study, we would like to characterize the molecular profile of breast cancer among Chinese women in Hong Kong and associate the molecular features with clinical and etiologic factors. An improved understanding of the inter-relationships among age, breast cancer subtypes, and race/ethnicity is critical for the development of targeted prevention and the best and most efficacious therapy.

Objectives: To assess the technical feasibility of 1) collecting fresh frozen tissues and fixed tissue blocks from breast cancer cases in Hong Kong, and 2) conducting tumor profiling analyses in the collected tissues.

Eligibility: Breast cancer cases who are participants in an ongoing breast cancer case control study among Hong Kong women (Night shift and breast cancer: a case-control study among Hong Kong women, led by Dr. Tse at Chinese University in Hong Kong) and who will receive surgery at the North District Hospital, HK, in 2013.

Design: In this feasibility study, we plan to collect fresh frozen and fixed tissues (tumor and adjacent normal) from approximately 100 breast cancer cases who have given consent to participate in our breast tissue collection pilot study. DNA and RNA will be extracted from frozen tumors and assessed for quality and yield. We will then conduct expression profiling analysis in a subset of cases (N approximately 10) to determine the quality of RNA in molecular profiling analysis. We will also determine whether there are enough epithelial benign and tumor tissues for the construction of tissue microarrays (TMAs). The results from this feasibility study will inform our decision on whether or not to pursue a large scale study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects who are participants in an ongoing breast cancer case-control study among Hong Kong women (Night shift and breast cancer: a case-control study among Hong Kong women, led by Dr. Tse at Chinese University in Hong Kong) and who will receive surgery at the North District Hospital, HK, age 18-100 years, inclusive.

EXCLUSION CRITERIA:

Males, non-Asians, and children under 18 years will be excluded.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female breast cancer patients identified from the Surgery or Oncology Departments of two hospitals in Hong Kong (North District Hospital and Yan Chai Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-06-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
To collect fresh frozen breast tissues and 500 formalin-fixed parafin-embedded (FFPE) tissue blocks from 500 Hong Kong breast cancer cases | 12/31/2018
  Breast Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Rose Yang, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- China (2):
  - North District Hospital, Hong Kong
  - Yan Chai Hospital, Hong Kong

REFERENCES:
- [Background] Sung H, Rosenberg PS, Chen WQ, Hartman M, Lim WY, Chia KS, Wai-Kong Mang O, Chiang CJ, Kang D, Ngan RK, Tse LA, Anderson WF, Yang XR. Female breast cancer incidence among Asian and Western populations: more similar than expected. J Natl Cancer Inst. 2015 Apr 13;107(7):djv107. doi: 10.1093/jnci/djv107. Print 2015 Jul. PMID 25868578
- [Background] Sung H, Rosenberg PS, Chen WQ, Hartman M, Lim WY, Chia KS, Wai-Kong Mang O, Tse L, Anderson WF, Yang XR. The impact of breast cancer-specific birth cohort effects among younger and older Chinese populations. Int J Cancer. 2016 Aug 1;139(3):527-34. doi: 10.1002/ijc.30095. Epub 2016 Apr 9. PMID 26992019
- [Background] Li M, Tse LA, Chan WC, Kwok CH, Leung SL, Wu C, Yu WC, Yu IT, Yu CH, Wang F, Sung H, Yang XR. Evaluation of breast cancer risk associated with tea consumption by menopausal and estrogen receptor status among Chinese women in Hong Kong. Cancer Epidemiol. 2016 Feb;40:73-8. doi: 10.1016/j.canep.2015.11.013. Epub 2015 Dec 8. PMID 26680603